CLINICAL TRIAL: NCT01600105
Title: Prospective Detection of Liver Fibrosis With MRI Compared to Fibroscan and Blood Tests
Brief Title: Detection of Liver Fibrosis With Magnetic Resonance Imaging (MRI)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bachir Taouli (Other)
Responsible Party: Sponsor-Investigator, Bachir Taouli, Associate Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GCO 09-1187
Record Dates: First submitted 2012-05-14; First posted 2012-05-16 (Estimated); Results first posted 2019-03-11 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-01

CONDITIONS: Chronic Liver Disease
Keywords: liver fibrosis; liver cirrhosis; chronic hepatitis; magnetic resonance imaging
MeSH Terms: conditions — Liver Cirrhosis; Hepatitis, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Perfusion MRI (Experimental): chronic liver disease who underwent/will undergo liver biopsy or will undergo liver transplant or liver resection as part of standard care during the previous 6 months.
  Interventions: Drug: Perfusion MRI

INTERVENTIONS:
Drug: Perfusion MRI — 1) Assess the role of a new FDA approved blood pool gadolinium contrast agent (gadofosveset trisodium, Ablavar, Lantheus) for the measurement of liver MR Perfusion, compared to extra-cellular contrast agents.
  Other Names: Dynamic contrast-enhanced MRI; Perfusion MRI (adofosveset trisodium, Ablavar, Lantheus)

SUMMARY:
Patients with chronic liver disease are at high risk of developing liver scarring (fibrosis), with ultimate risks of cirrhosis and liver cancer that may require liver transplant. The investigators would like to develop non invasive advanced Magnetic Resonance Imaging (MRI) techniques (MR diffusion, perfusion and elastography) to assess the degree of liver damage in patients with chronic liver disease. These techniques combined could reach high diagnostic performance for detection of liver fibrosis; and could decrease the number of liver biopsies, which have risks and sample only a small portion of the liver.

DETAILED DESCRIPTION:
Patients with chronic hepatitis have increased risks of liver damage, including fibrosis and cirrhosis, which may eventually lead to hepatocellular carcinoma and end-stage liver disease requiring liver transplantation. These diseases are/will be the source of enormous health care costs and morbidity/mortality in the US.

Most hepatologists still rely on liver biopsy findings in patients newly diagnosed with chronic hepatitis, which enables the assessment of liver damage (fibrosis and inflammation). Liver biopsy has limitations, including cost, invasiveness, poor patient acceptance, limited sampling, inter-observer variability and is difficult to repeat.

Non invasive tests to capture the extent of liver damage at a larger scale are urgently needed. These will gain more acceptance among patients and hepatologists.

In this proposal, the investigators would like to test and validate non invasive MRI methods based on advanced MR diffusion, perfusion and elastography techniques for the detection of fibrosis and cirrhosis in patients with chronic hepatitis. In order to improve the diagnostic performance of MRI, the investigators would like to build and validate a predictive model based on advanced functional MRI metrics (diffusion, perfusion and elastography). If validated, this novel non invasive algorithm will not only decreases the number of liver biopsies, but also enable earlier diagnosis of liver fibrosis when antiviral treatment is more effective, and enable a comprehensive evaluation of the liver (to assess for cirrhosis, portal hypertension and hepatocellular cancer).

This could significantly reduce the cost of care, could become a useful tool for testing new antifibrogenic and antiviral drugs in chronic viral hepatitis, and could be used to follow patients for detection of progression to cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Chronic liver disease (including viral hepatitis, alcoholic hepatitis, non alcoholic steatohepatitis, primary biliary cirrhosis, primary sclerosing cholangitis, etc..)
* 18 years of age and older
* Liver biopsy (percutaneous or transjugular or surgical) performed within 6 months, as part of routine clinical care.
* Liver transplant or liver resection performed within 6 months, as part of routine clinical care.
* Patient is able to give informed consent for this study and agrees to provide a blood sample

Control group

* Patients without history of liver disease and healthy volunteers
* 18 years of age and older
* Subject is able to give informed consent for this study and agrees to provide a blood sample

Exclusion Criteria:

* Age less than 18 years
* Unable or unwilling to give informed consent
* Contra-indications to MRI
* Electrical implants such as cardiac pacemakers or perfusion pumps
* Ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the eye, or steel implants
* Ferromagnetic objects such as jewelry or metal clips in clothing
* Pregnant subjects
* Pre-existing medical conditions including a likelihood of developing seizures or claustrophobic reactions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2010-10; Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bachir Taouli, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Result] Jajamovich GH, Dyvorne H, Donnerhack C, Taouli B. Quantitative liver MRI combining phase contrast imaging, elastography, and DWI: assessment of reproducibility and postprandial effect at 3.0 T. PLoS One. 2014 May 19;9(5):e97355. doi: 10.1371/journal.pone.0097355. eCollection 2014. PMID 24840288
- [Result] Dyvorne HA, Jajamovich GH, Bane O, Fiel MI, Chou H, Schiano TD, Dieterich D, Babb JS, Friedman SL, Taouli B. Prospective comparison of magnetic resonance imaging to transient elastography and serum markers for liver fibrosis detection. Liver Int. 2016 May;36(5):659-66. doi: 10.1111/liv.13058. Epub 2016 Feb 7. PMID 26744140
- [Result] Wagner M, Hectors S, Bane O, Gordic S, Kennedy P, Besa C, Schiano TD, Thung S, Fischman A, Taouli B. Noninvasive prediction of portal pressure with MR elastography and DCE-MRI of the liver and spleen: Preliminary results. J Magn Reson Imaging. 2018 Oct;48(4):1091-1103. doi: 10.1002/jmri.26026. Epub 2018 Apr 11. PMID 29638020
- [Derived] Jajamovich GH, Calcagno C, Dyvorne HA, Rusinek H, Taouli B. DCE-MRI of the liver: reconstruction of the arterial input function using a low dose pre-bolus contrast injection. PLoS One. 2014 Dec 29;9(12):e115667. doi: 10.1371/journal.pone.0115667. eCollection 2014. PMID 25546176

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in May 2010, with enrollment from October 2010 through February 2017. Patients were recruited from the Division of Liver Diseases or from the Surgical Oncology Clinic at Mount Sinai.
Groups:
- Chronic Liver Disease Patients: chronic liver disease who underwent/will undergo liver biopsy or will undergo liver transplant or liver resection as part of standard care during the previous 6 months.
  Sub Study I: Patients were enrolled in the study if they had a liver biopsy performed within 3 months of the MRI study or were diagnosed with liver cirrhosis based on imaging findings.
  Sub Study II: Patients with mixed etiology of liver fibrosis proven by biopsy, and/or liver cirrhosis.
  Sub study III: Patients with chronic liver disease who underwent invasive hepatic vein pressure gradient (HVPG) measurement
- Healthy Volunteers: Healthy Volunteer for Sub study I
Period: Total Participants
Arm/Group | Chronic Liver Disease Patients | Healthy Volunteers
Started | 255 | 21
Completed | 214 | 11
Not Completed | 41 | 10
Not completed — Withdrawal by Subject | 1 | 0
Not completed — No images in PACS | 10 | 0
Not completed — Insufficient image quality | 30 | 10
Period: Sub Study I
Arm/Group | Chronic Liver Disease Patients | Healthy Volunteers
Started | 19 | 21
Completed | 19 | 11
Not Completed | 0 | 10
Not completed — Insufficient image quality | 0 | 10
Period: Sub Study II
Arm/Group | Chronic Liver Disease Patients | Healthy Volunteers
Started | 65 | 0
Completed | 60 | 0
Not Completed | 5 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — No images in PACS | 1 | 0
Not completed — Insufficient image quality | 3 | 0
Period: Sub Study III
Arm/Group | Chronic Liver Disease Patients | Healthy Volunteers
Started | 39 | 0
Completed | 34 | 0
Not Completed | 5 | 0
Not completed — Insufficient image quality | 5 | 0
Period: Sub Study IV
Arm/Group | Chronic Liver Disease Patients | Healthy Volunteers
Started | 41 | 8
Completed | 41 | 8
Not Completed | 0 | 0
Period: Sub Study V
Arm/Group | Chronic Liver Disease Patients | Healthy Volunteers
Started | 52 | 0
Completed | 50 | 0
Not Completed | 2 | 0
Not completed — Poor Image Quality | 2 | 0

BASELINE CHARACTERISTICS:
Population: This is the overall participants who completed the study. Substudies were conducted with participants pulled from the overall enrollment. There was no overall study with outcome measures for the overall enrollment
Groups:
- Healthy Volunteers: Healthy Volunteers in Sub study I only
- Total: Total of all reporting groups
Arm/Group | Perfusion MRI | Healthy Volunteers | Total
Number analyzed (Participants) | 214 | 11 | 225
Age, Continuous [Mean (Full Range); unit: years] | 53.8 [19 to 82] | 30.6 [19 to 42] | 51.8 [19 to 82]
Age, Customized [Mean (Full Range); unit: years] — Participants for Sub Study I Population: 30 Participants in Sub Study I: 11 healthy volunteers and 19 patients
  years
    Sub Study I Chronic Hepatitis C patients: number analyzed (Participants) | 19 | 11 | 30
    Sub Study I Chronic Hepatitis C patients | 55.8 [34 to 68] | 30.6 [19 to 42] | 46.5 [19 to 68]
Age, Customized [Mean (Full Range); unit: years] — Sub-study II had 60 participants Population: Sub-Study II with 60 participants
  years
    Sub Study II: number analyzed (Participants) | 60 | 0 | 60
    Sub Study II | 55 [23 to 69] |  | 55 [23 to 69]
Age, Customized [Mean (Full Range); unit: years] — Sub-Study III 34 participants who underwent HVPG measurements Population: Sub-Study III 34 participants who underwent HVPG measurements
  years
    Sub Study III: number analyzed (Participants) | 34 | 0 | 34
    Sub Study III | 53 [26 to 74] |  | 53 [26 to 74]
Age, Customized [Mean (Full Range); unit: years] — Sub Study IV - participants who underwent MRE at 3.0T Population: Sub Study IV had 49 participants - 41 with chronic liver disease and 8 healthy volunteers
  years
    Sub Study IV: number analyzed (Participants) | 41 | 8 | 49
    Sub Study IV | 53 [21 to 70] | 29 [19 to 39] | 48 [19 to 70]
Age, Customized [Mean (Full Range); unit: years] — Sub Study V: Participants who underwent 4D flow MRI Population: Sub Study V had 52 participants
  years
    Sub Study V: number analyzed (Participants) | 52 | 0 | 52
    Sub Study V | 57 [22 to 82] |  | 57 [22 to 82]
Sex: Female, Male [Count of Participants; unit: Participants] — For overall participants that completed study Population: Participants who completed study
  Participants
    Female | 83 | 5 | 88
    Male | 131 | 6 | 137
Sex: Female, Male [Count of Participants; unit: Participants] — Sub-Study I - 30 Participants Population: 30 Participants in Sub Study I
  Participants
    Chronic Hepatitis C patients: number analyzed (Participants) | 19 | 11 | 30
    Chronic Hepatitis C patients: Female | 2 | 5 | 7
    Chronic Hepatitis C patients: Male | 17 | 6 | 23
Sex: Female, Male [Count of Participants; unit: Participants] — Sub-Study II with 60 participants Population: Sub-study II with 60 participants
  Participants
    number analyzed (Participants) | 60 | 0 | 60
    Female | 20 |  | 20
    Male | 40 |  | 40
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sub Study III had 34 participants
  Participants
    number analyzed (Participants) | 34 | 0 | 34
    Female | 18 |  | 18
    Male | 16 |  | 16
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sub Study IV had 49 participants
  Participants
    number analyzed (Participants) | 41 | 8 | 49
    Female | 18 | 5 | 23
    Male | 23 | 3 | 26
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sub Study V had 52 participants
  Participants
    number analyzed (Participants) | 52 | 0 | 52
    Female | 20 |  | 20
    Male | 32 |  | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Participants who completed study.
  Participants
    White | 105 | 3 | 108
    Asian | 31 | 1 | 32
    Black or African American | 20 | 5 | 25
    Hispanic | 38 | 2 | 40
    Unknown | 20 | 0 | 20

OUTCOME MEASURES:

1. Primary Outcome: PV Flow
Description: Sub-Study I Portal Venous Flow - forward flow during systole and early diastole, and flow reversal after atrial contraction.The average PV area was extracted, and PV flow was computed as the multiplication of area and velocity.
Time Frame: Fasting State Scan (an average of 15 min) and Postprandial State Scan (an average of 15 min)
Measure: Mean (Standard Deviation); unit: ml/s
Groups:
- Chronic Hep C Patients: chronic liver disease who underwent/will undergo liver biopsy or will undergo liver transplant or liver resection as part of standard care during the previous 6 months.
  Perfusion MRI: 1) Assess the role of a new FDA approved blood pool gadolinium contrast agent (gadofosveset trisodium, Ablavar, Lantheus) for the measurement of liver MR Perfusion, compared to extra-cellular contrast agents.
- Healthy Volunteers: No Hep C
Arm/Group | Chronic Hep C Patients | Healthy Volunteers
Number analyzed (Participants) | 19 | 11
ml/s
  Fasting | 16.0 (6.1) | 15.5 (4.2)
  Postprandial | 23.2 (8.5) | 27.1 (10.2)

2. Primary Outcome: PV Velocity
Description: Sub-Study I Portal Venous Flow Velocity - The mean velocity of the region of interest (ROI) was extracted for each one of the 25 phase images, and the time average was computed.
Time Frame: Fasting State Scan (an average of 15 min) and Postprandial State Scan (an average of 15 min)
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Chronic Hep C Patients | Healthy Volunteers
Number analyzed (Participants) | 19 | 11
cm/s
  Fasting | 10.5 (3.2) | 11.5 (2.8)
  Postprandial | 12.8 (4.6) | 14.4 (3.2)

3. Primary Outcome: LS-MRE for Sub-Study I
Description: Sub-Study I Liver stiffness (LS) measured by magnetic resonance elastography (MRE) in kilopascal (kPa). Liver stiffness is assessed by mathematical modeling of compression waves propagation in the liver, as measured from MRE images.
Time Frame: Fasting State Scan (an average of 15 min) and Postprandial State Scan (an average of 15 min)
Population: Sub Study I with 30 participants. The method failed in 3 of the patients, so no usable LS-MRE data was generated. 27 patients had usable data for PV flow and velocity, so they were included in the study.
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Chronic Hep C Patients | Healthy Volunteers
Number analyzed (Participants) | 19 | 11
kPa
  Fasting: number analyzed (Participants) | 16 | 11
  Fasting | 4.9 (1.4) | 1.8 (0.2)
  Postprandial | 5.0 (1.2) | 2.0 (0.2)

4. Primary Outcome: True Diffusion Parameter (D)
Description: Sub-Study II True Diffusion Parameter - D- describes water diffusion in tissue independently from the effects of capillary perfusion; it is obtained from bi-exponential fitting of MRI diffusion signal acquired over a range of high and low diffusion-weighting factors (b-values)
  Fibrosis State/Score:
  F0-F2 - no signs of fibrosis to minimal fibrosis F3-F4 - fibrosis has spread and has connected to other areas on the liver that contain fibrosis or presence of cirrhosis
Time Frame: Fasting State Multiparametric MRI Scan (an average of 60 min) Scan
Population: 3 participants with scans not evaluable
Measure: Mean (Standard Deviation); unit: 10^-3 mm^2/s
Arm/Group | Perfusion MRI
Number analyzed (Participants) | 57
10^-3 mm^2/s
  F0-F2: number analyzed (Participants) | 31
  F0-F2 | 1.06 (0.21)
  F3-F4: number analyzed (Participants) | 26
  F3-F4 | 0.94 (0.16)

5. Primary Outcome: LS-MRE Fibrosis State for Sub Study II
Description: Sub-Study II Liver stiffness (LS) measured by magnetic resonance elastography (MRE) in kilopascal (kPa). Liver stiffness is assessed by mathematical modeling of compression waves propagation in the liver, as measured from MRE images.
  Fibrosis State/Score:
  F0-F2 - no signs of fibrosis to minimal fibrosis F3-F4 - fibrosis has spread and has connected to other areas on the liver that contain fibrosis or presence of cirrhosis
Time Frame: Fasting State Multiparametric MRI Scan (an average of 60 min)
Population: Only 38 participants had suitable MRE quality for analysis.
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Perfusion MRI
Number analyzed (Participants) | 38
kPa
  F0-F2: number analyzed (Participants) | 24
  F0-F2 | 2.88 (0.91)
  F3-F4: number analyzed (Participants) | 14
  F3-F4 | 5.16 (0.95)

6. Primary Outcome: LS-TE
Description: Sub-Study II Liver Stiffness with transient elastography (TE) (LS-TE) - a non-invasive modality of liver fibrosis detection: a shear wave is sent into the liver through a small transducer attached to an ultrasound probe, and the velocity of the wave is measured as it passes through the liver; shear wave velocity is then converted to stiffness, measured in kilopascals (kPa)
  Fibrosis State/Score:
  F0-F2 - no signs of fibrosis to minimal fibrosis F3-F4 - fibrosis has spread and has connected to other areas on the liver that contain fibrosis or presence of cirrhosis
Time Frame: Fasting transient elastography, average duration 10 min
Population: Only 46 participants had suitable TE quality for analysis.
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Perfusion MRI
Number analyzed (Participants) | 46
kPa
  F0-F2: number analyzed (Participants) | 23
  F0-F2 | 9.55 (6.85)
  F3-F4: number analyzed (Participants) | 23
  F3-F4 | 21.44 (17.86)

7. Primary Outcome: MTT
Description: Sub-Study II Mean Transit Time (MTT) - Liver Mean Transit Time of Contrast Agent through the tissue of interest from Dynamic Contrast Enhanced MRI
  Fibrosis State/Score:
  F0-F2 - no signs of fibrosis to minimal fibrosis F3-F4 - fibrosis has spread and has connected to other areas on the liver that contain fibrosis or presence of cirrhosis
Time Frame: Fasting State Multiparametric MRI Scan (an average of 60 min)
Population: Only 50 participants had suitable quality MRI for analysis
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Perfusion MRI
Number analyzed (Participants) | 50
seconds
  F0-F2: number analyzed (Participants) | 25
  F0-F2 | 11.6 (8.1)
  F3-F4: number analyzed (Participants) | 25
  F3-F4 | 18.8 (9.1)

8. Secondary Outcome: Liver Upslope From DCE-MRI
Description: Sub-Study III Liver Upslope of MRI signal is defined as peak concentration to the time to reach peak concentration of gadolinium contrast agent in the liver tissue of interest, derived from dynamic contrast-enhanced MRI (DCE-MRI.
  Portal hypertension (PH), defined by hepatic venous pressure gradient (HVPG) ≥5 mmHg Clinically Significant Portal hypertension (CSPH), defined by hepatic venous pressure gradient (HVPG) ≥10 mmHg
Time Frame: Fasting State Multiparametric MRI Scan (an average of 60 min)
Population: Among the 34 patients, 2 patients did not have DCE-MRI acquisition due to chronic renal insufficiency, 4 patients had non-usable DCE-MRI data because of major artifacts.
Measure: Median (Standard Deviation); unit: mmol/(L.s))
Arm/Group | Perfusion MRI
Number analyzed (Participants) | 28
mmol/(L.s))
  HVPG <5mmHg: number analyzed (Participants) | 12
  HVPG <5mmHg | 0.011 (0.011)
  HVPG>=5mmHg: number analyzed (Participants) | 16
  HVPG>=5mmHg | 0.0007 (0.0007)
  HPVG<10mmHg: number analyzed (Participants) | 20
  HPVG<10mmHg | 0.011 (0.007)
  HPVG>=10mmHg: number analyzed (Participants) | 8
  HPVG>=10mmHg | 0.0006 (0.004)

9. Secondary Outcome: Liver Time to Peak (TTP) for PH
Description: Sub-Study III Liver Time to Peak (TTP) is defined as the time in seconds to reach peak concentration of gadolinium contrast agent in the liver tissue of interest, derived from dynamic contrast-enhanced MRI (DCE-MRI) Portal hypertension (PH), defined by hepatic venous pressure gradient (HVPG) ≥5 mmHg Clinically Significant Portal Hypertension is defined as an HVPG ≥10 mmHg
Time Frame: Fasting State Multiparametric MRI Scan (an average of 60 min)
Population: as for outcome 8
Measure: Median (Standard Deviation); unit: seconds
Arm/Group | Perfusion MRI
Number analyzed (Participants) | 28
seconds
  HVPG<5mmHg: number analyzed (Participants) | 12
  HVPG<5mmHg | 40.99 (22.20)
  HVPG>=5mmHg: number analyzed (Participants) | 16
  HVPG>=5mmHg | 53.02 (31.8)
  HVPG<10mmHg: number analyzed (Participants) | 20
  HVPG<10mmHg | 41.47 (25.76)
  HVPG>=10mmHg: number analyzed (Participants) | 8
  HVPG>=10mmHg | 69.45 (41.98)

10. Secondary Outcome: LS-MRE Portal Hypertension for Sub Study III
Description: Sub-Study III Liver stiffness (LS) measured by magnetic resonance elastography (MRE) in kilopascal (kPa). Liver stiffness is assessed by mathematical modeling of compression waves propagation in the liver, as measured from MRE images.
  Portal Hypertension is defined as an HVPG ≥5 mmHg Clinically Significant Portal hypertension (CSPH), defined by hepatic venous pressure gradient (HVPG) ≥10 mmHg
Time Frame: Fasting State Multiparametric MRI Scan (an average of 60 min)
Population: MRE was successful for liver stiffness measurements in 31 participants of the 34
Measure: Median (Standard Deviation); unit: kPa
Arm/Group | Perfusion MRI
Number analyzed (Participants) | 31
kPa
  HVPG<5mmHg: number analyzed (Participants) | 12
  HVPG<5mmHg | 2.31 (2.8)
  HVPG>=5mmHg: number analyzed (Participants) | 19
  HVPG>=5mmHg | 5.14 (2.57)
  HVPG<10mmHg: number analyzed (Participants) | 22
  HVPG<10mmHg | 3.88 (3.16)
  HVPG>=10mmHg: number analyzed (Participants) | 9
  HVPG>=10mmHg | 5.86 (6.71)

11. Secondary Outcome: Spleen Volume
Description: Sub-Study III Portal Hypertension is defined as an HVPG ≥5 mmHg
Time Frame: Fasting State Multiparametric MRI Scan (an average of 60 min)
Population: Sub Study III with 34 participants
Measure: Median (Standard Deviation); unit: cm^3
Arm/Group | Perfusion MRI
Number analyzed (Participants) | 34
cm^3
  HVPG<5mmHg: number analyzed (Participants) | 12
  HVPG<5mmHg | 246 (252)
  HVPG>=5mmHg: number analyzed (Participants) | 22
  HVPG>=5mmHg | 441 (629)

12. Secondary Outcome: Spleen Caudocranial Diameter
Description: Sub-Study III Portal Hypertension is defined as an HVPG ≥5 mmHg
Time Frame: Fasting State Multiparametric MRI Scan (an average of 60 min)
Population: Sub Study III with 34 participants
Measure: Median (Standard Deviation); unit: cm
Arm/Group | Perfusion MRI
Number analyzed (Participants) | 34
cm
  HVPG<5mmHg: number analyzed (Participants) | 12
  HVPG<5mmHg | 11.6 (2.8)
  HVPG>=5mmHg: number analyzed (Participants) | 22
  HVPG>=5mmHg | 14.0 (4.8)

13. Secondary Outcome: PH Imaging Score
Description: Sub-Study III Portal Hypertension imaging composite score (based on the presence of varices, spleen size, presence of ascites). The imaging score is based on the number of variceal sites (0: absence of varices, 1: one variceal site, 2: two variceal sites, and 3: 3 or more variceal sites), volume of ascites (0: no ascites, 1: minimal perihepatic and perisplenic fluid, 2: intraperitoneal fluid without marked abdominal wall distension, and 3: fluid causing marked abdominal wall distension), and maximum craniocaudal diameter of the spleen (0: size less than 13 cm, 1: size between 13 and 15 cm, 2: size between 15 and 20 cm, and 3: size greater than 20 cm). Score from 0 to 9, with higher score indicating worse disease.
  Portal Hypertension is defined as an HVPG ≥5 mmHg Clinically Significant Portal hypertension (CSPH), defined by hepatic venous pressure gradient (HVPG) ≥10 mmHg
Time Frame: Fasting State Multiparametric MRI Scan (an average of 60 min)
Population: Sub Study III with 34 participants
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Perfusion MRI
Number analyzed (Participants) | 34
score on a scale
  HVPG<5mmHg: number analyzed (Participants) | 12
  HVPG<5mmHg | 0 (1)
  HVPG>=5mmHg: number analyzed (Participants) | 22
  HVPG>=5mmHg | 2 (5.25)
  HVPG<10: number analyzed (Participants) | 25
  HVPG<10 | 1 (1.5)
  HVPG>=10: number analyzed (Participants) | 9
  HVPG>=10 | 4 (4.5)

14. Secondary Outcome: LSLU
Description: Sub-Study III Liver Stiffness to Liver Upslope ratio (LSLU) Portal Hypertension is defined as an HVPG ≥5 mmHg Clinically Significant Portal hypertension (CSPH), defined by hepatic venous pressure gradient (HVPG) ≥10 mmHg
Time Frame: Fasting State Multiparametric MRI Scan (an average of 60 min)
Population: 31 of the 34 participants had LS-MRE and 28 of the 34 participants had Liver Upslope measurement from DCE-MRI
Measure: Median (Standard Deviation); unit: kPa*s*L/mmol
Arm/Group | Perfusion MRI
Number analyzed (Participants) | 28
kPa*s*L/mmol
  HVPG<5mmHg: number analyzed (Participants) | 12
  HVPG<5mmHg | 192.72 (195.65)
  HVPG>=5mmHg: number analyzed (Participants) | 16
  HVPG>=5mmHg | 830.28 (971.68)
  HVPG<10mmHg: number analyzed (Participants) | 20
  HVPG<10mmHg | 363.68 (855.01)
  HVPG>10mmHg: number analyzed (Participants) | 8
  HVPG>10mmHg | 871.82 (1354.31)

15. Secondary Outcome: Liver DV
Description: Sub Study III Liver Distribution Volume (DV) is the distribution volume of contrast agent in the tissue of interest defined as a percentage ratio of gadolinium material volume to the volume of the liver tissue of interest, as derived from DCE-MRI; in the case of a contrast agent with extracellular distribution, DV measures the intravascular and extravascular-extracellular volume.
  Clinically Significant Portal hypertension (CSPH), defined by hepatic venous pressure gradient (HVPG) ≥10 mmHg
Time Frame: Fasting State Multiparametric MRI Scan (an average of 60 min)
Population: as for outcome 8
Measure: Median (Standard Deviation); unit: percentage of liver volume
Arm/Group | Perfusion MRI
Number analyzed (Participants) | 28
percentage of liver volume
  HVPG<10mmHg: number analyzed (Participants) | 20
  HVPG<10mmHg | 47.28 (24.29)
  HVPG>=10mmHg: number analyzed (Participants) | 8
  HVPG>=10mmHg | 77.25 (111.01)

16. Secondary Outcome: Spleen TTP
Description: Sub Study III Spleen Time To Peak (TTP) - time to reach peak gadolinium concentration in spleen tissue of interest, derived from DCE-MRI.
  Clinically Significant Portal hypertension (CSPH), defined by hepatic venous pressure gradient (HVPG) ≥10 mmHg
Time Frame: Fasting State Multiparametric MRI Scan (an average of 60 min)
Population: as for outcome 8
Measure: Median (Standard Deviation); unit: seconds
Arm/Group | Perfusion MRI
Number analyzed (Participants) | 28
seconds
  HVPG<10mmHg: number analyzed (Participants) | 20
  HVPG<10mmHg | 15.46 (16.65)
  HVPG>=10mmHg: number analyzed (Participants) | 8
  HVPG>=10mmHg | 44.90 (40.69)

ADVERSE EVENTS:
Time Frame: 6 years
Groups:
- Sub Study 1 Chronic Hep C Patients: Quantitative Liver MRI Combining Phase Contrast Imaging, Elastography, and DWI: Assessment of Reproducibility and Postprandial Effect Description: Patients with liver disease who had portal vein (PV) flow parameters measured with phase contrast (PC) imaging, liver diffusion parameters measured with multiple b value diffusion-weighted imaging (DWI) and liver stiffness (LS) measured with MR elastography (MRE) in fasting conditions and after a meal challenge.
- Sub Study 1 Health Volunteers: Quantitative Liver MRI Combining Phase Contrast Imaging, Elastography, and DWI: Assessment of Reproducibility and Postprandial Effect Description: Healthy volunteers who had portal vein (PV) flow parameters measured with phase contrast (PC) imaging, liver diffusion parameters measured with multiple b value diffusion-weighted imaging (DWI) and liver stiffness (LS) measured with MR elastography (MRE) in fasting conditions and after a meal challenge.
- Sub Study II: Arm/Group Title: Prospective Comparison of Magnetic Resonance Imaging to Transient Elastography and Serum Markers for Liver Fibrosis Detection Description: Chronic liver disease patients who underwent a multiparametric magnetic resonance imaging (MRI) protocol including diffusion�\weighted imaging (DWI), dynamic contrast�\enhanced (DCE)�\MRI and magnetic resonance elastography (MRE) in comparison with transient elastography (TE) for liver fibrosis detection.
- Sub Study III: Noninvasive Prediction of Portal Pressure with MR Elastography and DCE�\MRI of the Liver and Spleen Description: Chronic liver disease patients who underwent HVPG measurement, MR elastography (MRE) and dynamic contrast�\enhanced MRI (DCE�\MRI) of the liver and spleen
- Total Participants of the Substudies: Total participants of Sub Study 1, Sub Study II, and Sub Study III
Arm/Group | Sub Study 1 Chronic Hep C Patients | Sub Study 1 Health Volunteers | Sub Study II | Sub Study III | Total Participants of the Substudies
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/11 | 0/60 | 0/34 | 0/124
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/11 | 0/60 | 0/34 | 0/124
Other Adverse Events (participants affected / at risk) | 0/19 | 0/11 | 2/60 | 0/34 | 2/124
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sub Study 1 Chronic Hep C Patients (N=19) | Sub Study 1 Health Volunteers (N=11) | Sub Study II (N=60) | Sub Study III (N=34) | Total Participants of the Substudies (N=124)
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Fainting (Nervous system disorders) | 0 | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-16): https://cdn.clinicaltrials.gov/large-docs/05/NCT01600105/Prot_SAP_000.pdf